CLINICAL TRIAL: NCT01045174
Title: A Randomized Controlled Trial Comparing the Effectiveness of a Breath-Actuated Nebulizer Device Versus a Conventional Continuous-Output Nebulizer in Treating Pediatric Asthma Patients in the Emergency Department
Brief Title: Breath-Actuated Nebulizer Versus Conventional Continuous-Output Nebulizer in Pediatric Asthma Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in availability of study investigators
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jerri A. Rose, M.D., University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UH IRB # 09-08-06
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Asthma; Pediatric; Emergency department; Nebulizer
MeSH Terms: conditions — Asthma; Emergencies | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breath-Actuated Nebulizer (Active Comparator): Participants are randomly assigned to receive bronchodilator treatments for asthma according to the standard of care using either a breath-actuated nebulizer device or a conventional continuous-output nebulizer.
  Interventions: Device: Nebulizer (breath-actuated versus conventional continuous-output)
- Conventional continuous-ouput nebulizer (Active Comparator): Participants are randomly assigned to receive bronchodilator treatments for asthma according to the standard of care using either a breath-actuated nebulizer device or a conventional continuous-output nebulizer
  Interventions: Device: Nebulizer (breath-actuated versus conventional continuous-output)

INTERVENTIONS:
Device: Nebulizer (breath-actuated versus conventional continuous-output) — Participants are randomly assigned to receive bronchodilator treatments for asthma according to the standard of care using either a breath-actuated nebulizer device or a conventional continuous-output nebulizer. Standard unit doses of albuterol/ipratropium bromide or albuterol are used in both devices.

SUMMARY:
A Breath-Actuated Nebulizer is a newer type of nebulizer device that creates aerosol only when a patient is inhaling, rather than creating aerosol continuously. It is thought that breath-actuated nebulizer devices may deliver asthma rescue medications to patients' lungs more effectively and therefore lead them to recover from asthma attacks faster than conventional continuous-output nebulizer devices. This study compares outcomes including hospital admission rates, number of nebulized treatments required, and patient/family satisfaction when a breath-actuated nebulizer device versus a conventional continuous-output nebulizer is used to deliver asthma medications to pediatric asthma patients in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* children 1-17 years old with known history of asthma
* children must be presenting to the emergency department for treatment of acute asthma
* children must qualify to be treated for acute asthma according to an existing standardized asthma care algorithm

Exclusion Criteria:

* concomitant chronic respiratory or cardiac disease such as cystic fibrosis, congenital heart disease, or bronchopulmonary dysplasia
* no prior history of asthma
* pregnancy
* reported history of drug allergy to albuterol or ipratropium bromide
* previous participation in the study within the preceding three weeks
* vital sign instability/need for immediate emergency intervention to prevent clinical deterioration

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerri A Rose, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Rainbow Babies and Children's Hospital/University Hospitals of Cleveland Pediatric Emergency Department, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants recruited from eligible children who presented to a pediatric emergency department at the single study site with acute asthma exacerbation/status asthmaticus. Recruitment for this study is now closed.
Pre-assignment Details: 180 participants were enrolled in the study. No enrolled participants were excluded from the study before assignment to groups.
Groups:
- Breath-Actuated Nebulizer: Participants randomly assigned to receive bronchodilator treatments for asthma according to the standard of care using either a breath-actuated nebulizer device or a conventional continuous-output nebulizer.
  Nebulizer (breath-actuated versus conventional continuous-output): Participants randomly assigned to receive bronchodilator treatments for asthma according to the standard of care using either a breath-actuated nebulizer device or a conventional continuous-output nebulizer. Standard unit doses of albuterol/ipratropium bromide or albuterol used in both devices.
- Conventional Continuous-ouput Nebulizer: Participants randomly assigned to receive bronchodilator treatments for asthma according to the standard of care using either a breath-actuated nebulizer device or a conventional continuous-output nebulizer
  Nebulizer (breath-actuated versus conventional continuous-output): Participants randomly assigned to receive bronchodilator treatments for asthma according to the standard of care using either a breath-actuated nebulizer device or a conventional continuous-output nebulizer. Standard unit doses of albuterol/ipratropium bromide or albuterol used in both devices.
Period: Overall Study
Arm/Group | Breath-Actuated Nebulizer | Conventional Continuous-ouput Nebulizer
Started | 90 | 90
Completed | 90 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breath-Actuated Nebulizer | Conventional Continuous-ouput Nebulizer | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 90 | 90 | 180
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 6.6 [2 to 17] | 6.7 [2 to 17] | 6.65 [2 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 44 | 90
  Male | 44 | 46 | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 90 | 90 | 180

OUTCOME MEASURES:

1. Primary Outcome: Rate of Admission to Hospital for Asthma Exacerbation
Description: Number (and percentage) of children in each study group requiring admission to the hospital for asthma exacerbation/status asthmaticus from the Pediatric Emergency Department (as opposed to being discharged to home)
Time Frame: 24 hours (whether patient is admitted after presenting to emergency department for asthma or discharged home)
Measure: Count of Participants; unit: Participants
Arm/Group | Breath-Actuated Nebulizer | Conventional Continuous-ouput Nebulizer
Number analyzed (Participants) | 90 | 90
Participants | 33 | 44

2. Secondary Outcome: Length of Stay in the Emergency Department After Presenting for Asthma Exacerbation
Description: Length of stay in the emergency department measured in minutes; up to 400 minutes measured
Time Frame: only measures length of stay in emergency department on date of presentation
Measure: Mean (Full Range); unit: minutes
Arm/Group | Breath-Actuated Nebulizer | Conventional Continuous-ouput Nebulizer
Number analyzed (Participants) | 90 | 90
minutes | 162 [90 to 375] | 178 [94 to 300]

3. Secondary Outcome: Patient's Satisfaction With Using Assigned Nebulizer (as Assessed by Brief Survey)
Description: Percentage of patients (or caregivers of younger children) who "agreed" or "strongly agreed" on a brief survey (using a 5-point Likert scale) that they would feel comfortable with using the same nebulizer device to take asthma treatments in the future. Likert-type scale was used, on which score of 1=strongly disagree, 2=disagree, 3=neither agree nor disagree (or unsure), 4=agree, and 5=strongly agree.
Time Frame: within time frame of emergency department stay (up to 400 minutes from initial presentation to pediatric ED)
Measure: Count of Participants; unit: Participants
Arm/Group | Breath-Actuated Nebulizer | Conventional Continuous-ouput Nebulizer
Number analyzed (Participants) | 90 | 90
Participants | 76 | 55

4. Secondary Outcome: Difficulty (if Any) Encountered by Patients With Using Assigned Nebulizer Device
Time Frame: number of children who had difficulty using assigned nebulizer device during the timeframe of the ED visit during which the study nebulizer was used. Timeframe for outcome measure was length of single emergency department visit, up to 400 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Breath-Actuated Nebulizer | Conventional Continuous-ouput Nebulizer
Number analyzed (Participants) | 90 | 90
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Breath-Actuated Nebulizer | Conventional Continuous-ouput Nebulizer
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No